CLINICAL TRIAL: NCT03748004
Title: Optimizing the Employment Outcomes for People Living in the Downtown Eastside
Brief Title: IPS/Peer Support Intervention in the DTES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Ministry of Social Development and Poverty Reduction, British Columbia (Other)
Responsible Party: Principal Investigator, Skye Barbic, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H18-02740
Record Dates: First submitted 2018-10-11; First posted 2018-11-20 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Behavior, Adaptive; Mental Illness; Substance Use
Keywords: Homeless; Employment
MeSH Terms: conditions — Behavior; Mental Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: 72 clients receiving primary care services from one DTES clinical site who are employment ready will be randomly assigned to IPS and Peer Support (experimental group) or WorkBC (control group).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults living in the DTES (Experimental): 36 out of the 72 recruited participants who live in the DTES will be randomly assigned to the intervention group (IPS & Peer Support). The IPS and Peer Support will actively work and support with each of the 36 participants in seeking employment and education for 16 weeks. IPS/SP will help participants identify their employment and educational goals, identify potential employers, help prepare their resumes and for interviews, and provide ongoing support during the 16 weeks.
  36 out of the 72 participants who live in the DTES will be randomly assigned to the control group (WorkBC). Participants will be provided with WorkBC employment services.
  Interventions: Behavioral: IPS/SP
- Individuals 19 yrs or older settled in DTES (Placebo Comparator): 36 out of the 72 recruited participants who live in the DTES will be randomly assigned to the intervention group (IPS & Peer Support). The IPS and Peer Support will actively work and support with each of the 36 participants in seeking employment and education for 16 weeks. IPS/SP will help participants identify their employment and educational goals, identify potential employers, help prepare their resumes and for interviews, and provide ongoing support during the 16 weeks.
  36 out of the 72 participants who live in the DTES will be randomly assigned to the control group (WorkBC). Participants will be provided with WorkBC employment services.
  Interventions: Behavioral: WorkBC

INTERVENTIONS:
Behavioral: IPS/SP — The 72 recruited clients receiving primary care services from one DTES clinical site who are employment ready will be randomly assigned to IPS and Peer Support (experimental group) or WorkBC control group
  Arms: Adults living in the DTES
Behavioral: WorkBC — 36 out of the 72 participants who live in the DTES will be randomly assigned to the control group (WorkBC). Participants will be provided with WorkBC employment services.
  Arms: Individuals 19 yrs or older settled in DTES

SUMMARY:
Individual placement support (IPS) is an evidence-based supported employment model for people with severe mental illness, designed to achieve employment in mainstream competitive jobs, either part-time or full-time. The aim of this study is to assess the (i) effectiveness of embedding the (IPS)/Peer Support intervention as part of the primary care centre in securing employment of adults living in the downtown eastside in comparison to the usual treatment WorkBC (control group). (ii) effectiveness of IPS/Peer Support versus the usual treatment (WorkBC) in improving mental illness, quality of life and personal recovery through participation in employment.

DETAILED DESCRIPTION:
This 18-month mixed methods study consists of an effectiveness multi-site randomized controlled trial of the IPS/peer support intervention plus an embedded qualitative exploration of participants' experiences. All clients receiving primary care services from one DTES clinical site who are employment ready and are not receiving mental health services will be randomly assigned to IPS & Peer Support (experimental group) or WorkBC (control group). Clients are required to participate in the intervention for 16 weeks and will be assessed at baseline, 1-, 3-, and 6-months post study intervention start-date for both groups. Assessments will include the 5 questionnaires administered at baseline which cover the following: Employment Quality, Employment Sustainability, Education Quality and Quantity, Quality of Life, Community Engagement and Clinical significant levels of depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 19 and over, accessing primary care services at the primary care centre listed in this study (CH Pender Community Health Centre)
* At least one visit to VCH Pender Community Health Centre
* Currently unemployed and not in school or post-secondary training.
* Able to provide informed consent and fluent in English (intervention is currently offered in English only).
* Not hospitalized at the time of recruitment.

Exclusion Criteria:

• Adults, age 19 and over who have access to mental health services

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Securing employment | 18 months
  RC will follow-up with all recruited clients who get employed through the IPS/Peer Support intervention and the WorkBC control group.

SECONDARY OUTCOMES:
"PHQ-9" Questionnaire to measures level of depression | 18 months
  Participants will answer the questions on this questionnaire using a likert scale. A scoring system will calculate the final total number and we will assess mean change from the baseline. The minimum score is 0/27 and the maximum score is 27
"GAD7" questionnaire to measure general anxiety disorder | 18 months
  Participants will answer the questions on this questionnaire using a likert scale. A scoring system will calculate the final total number and we will assess mean change from the baseline. The minimum score is 0/21. The maximum score is 21.
"C-PROM" questionnaire to measure Personal Recovery | 18 months
  Participants will answer the questions on this questionnaire using a likert scale. A scoring system will calculate the final total number and we will assess mean change from the baseline. Minimum score is 0/120. Maximum score is 120
"REQOL" questionnaire measures Recovery Quality of Life | 18 months
  Participants will answer the questions on this questionnaire using a likert scale. A scoring system will calculate the final total number and we will assess mean change from the baseline. Minimum score is 0/64. Maximum score 64.
"SWL" questionnaire measures satisfaction with life | 18 months
  Participants will answer the questions on this questionnaire using a likert scale. A scoring system will calculate the final total number and we will assess mean change from the baseline. Minimum score is 5/35. Maximum score is 35.

CONTACTS AND LOCATIONS:
Overall Officials: Skye Barbic, PhD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Downtown Community Health Center, Vancouver, British Columbia
  - Heatley Community Health Clinic, Vancouver, British Columbia
  - Pender Community Health Clinic, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No
It is a pilot study (early phase)

REFERENCES:
- [Background] Sveinsdottir V, Lovvik C, Fyhn T, Monstad K, Ludvigsen K, Overland S, Reme SE. Protocol for the effect evaluation of Individual Placement and Support (IPS): a randomized controlled multicenter trial of IPS versus treatment as usual for patients with moderate to severe mental illness in Norway. BMC Psychiatry. 2014 Nov 18;14:307. doi: 10.1186/s12888-014-0307-7. PMID 25403470
- [Background] Campbell K, Bond GR, Drake RE. Who benefits from supported employment: a meta-analytic study. Schizophr Bull. 2011 Mar;37(2):370-80. doi: 10.1093/schbul/sbp066. Epub 2009 Aug 6. PMID 19661196
- [Background] Latimer E, Lecomte T. [Individual Placement Support (IPS) for people with severe mental disorders : An approach to favor in Quebec?]. Sante Ment Que. 2002;27(1):241-67. French. PMID 18253627
- [Background] Bond GR, Drake RE. Making the case for IPS supported employment. Adm Policy Ment Health. 2014 Jan;41(1):69-73. doi: 10.1007/s10488-012-0444-6. PMID 23161326